CLINICAL TRIAL: NCT05785676
Title: Study of ALN's OATF Vena Cava Filter
Brief Title: ALN OATF Vena Cava Filter
Acronym: CONFIAL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Aln2b SARL (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP220570; 2022-A00915-38 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2023-03-09; First posted 2023-03-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Embolism
Keywords: Vena Cava Filter
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vena Cava Filter: Participants implanted with the vena cava filter OATF (ALN)
  Interventions: Device: Filter implantation

INTERVENTIONS:
Device: Filter implantation — Implantation of OATF ALN vena cava filter

SUMMARY:
Migration of a thrombus in the pulmonary circulation is the leading cause of pulmonary embolism (PE). It can be prevented mechanically by implanting a vena cava filter (VCF) in the inferior vena cava. The implation of a VCF is indicated for patients with acute PE and a contraindication to anticoagulation, with an acute deep vein thrombosis (DVT) without PE and a contraindication to anticoagulation or with acute venous thromboembolism (less than 3 months) in whom an interventional gesture at hemorrhagic and thromboembolic risk contraindicates anticoagulation.

The purpose of this study is to describe the rates of implantation, removal and complications associated with the use of the optional ALN OATF VCF in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with an ALN OATF VCF
* Patient informed

Exclusion Criteria:

* Minor patient
* Adult patient under a legal protection measure
* Pregnant, parturient or breastfeeding women
* Patient who refused to participate
* Patient who cannot or does not wish to be followed by the Interventional Radiology Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring a vena cave filter
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Filter implantation | day 0
  Rate of technical success of filter implantation

SECONDARY OUTCOMES:
Filter removal | up to 1 year
  Rate of filter removal

CONTACTS AND LOCATIONS:
Overall Officials: Olivier PELLERIN, MD - PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - Hôpital Européen Georges-Pompidou Paris, France, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).